CLINICAL TRIAL: NCT02169856
Title: A Randomized Controlled Trial: Role of EFTs (Emotional Freedom Techniques) in Reducing Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy.
Brief Title: Role of Emotional Freedom Techniques in Reducing Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Acronym: EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Dr.Fazal hussain Shah, Resident Surgery, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2014-06-09; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Cholecystectomy; Laparoscopic; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): control group was not given any EFTs (emotional freedom techniques) therapy for postoperative nausea and vomiting.
  Following medications were given to both groups. details are in respective interventions.
  Tab. Midazolam 7.5 mg Inj. Midazolam IV 0.7 mg/kg inj. propofol (2.5 mg/kg) inj. atracuium (0.5 mg/kg). sevoflurane (2.5 vol %) oxygen in air mixture (0.50 ratio) Inj. Cefuroxime 1.5 gm. IV Inj. Ketorolac 30mg IV Inj. Zantac 50 mg IV inj. Metoclopramide 10mg IV
  Interventions: Drug: Tab. Midazolam 7.5 mg; Drug: Inj. Midazolam 0.7mg/kg; Drug: Inj. Propofol 2.5mg/kg; Drug: Inj. Atracurium 0.5 mg/kg; Drug: Sevoflurane 2.5 vol %; Drug: Inj. Cefuroxime 1.5 g IV; Drug: Drug: Inj. Ketorolac 30 mg IV; Drug: Inj. Zantac 50mg IV
- EFTs study group (Experimental): EFTs (emotional freedom techniques) was applied to the patietns. one session of 5 to 10 min at 6 hours postoperatively.
  Following medications were given to both groups. details are in respective interventions.
  Tab. Midazolam 7.5 mg Inj. Midazolam IV 0.7 mg/kg inj. propofol (2.5 mg/kg) inj. atracuium (0.5 mg/kg). sevoflurane (2.5 vol %) oxygen in air mixture (0.50 ratio) Inj. Cefuroxime 1.5 gm. IV Inj. Ketorolac 30mg IV Inj. Zantac 50 mg IV inj. Metoclopramide 10mg IV
  Interventions: Behavioral: EFTs (emotional freedom techniques); Drug: Tab. Midazolam 7.5 mg; Drug: Inj. Midazolam 0.7mg/kg; Drug: Inj. Propofol 2.5mg/kg; Drug: Inj. Atracurium 0.5 mg/kg; Drug: Sevoflurane 2.5 vol %; Drug: Inj. Cefuroxime 1.5 g IV; Drug: Drug: Inj. Ketorolac 30 mg IV; Drug: Inj. Zantac 50mg IV

INTERVENTIONS:
Behavioral: EFTs (emotional freedom techniques) — The Emotional Freedom Techniques (EFTs) which has been pioneered by Gary Craig is a form of alternate medicine which works by tapping on body energy meridian points. Unlike drugs the EFTs has no side effects too
  Other Names: EFTs by garry craig
  Arms: EFTs study group
Drug: Tab. Midazolam 7.5 mg — Tab. Midazolam 7.5 mg will be given to all patients at night before surgery.
  Other Names: Tab. Doramicum
Drug: Inj. Midazolam 0.7mg/kg — Inj . Midazolam 0.7 mg/kg given as premedication 45 min before surgery.
  Other Names: inj. Doramicum
Drug: Inj. Propofol 2.5mg/kg — It was given to induce anesthesia after 3 min of pre oxygenation.
Drug: Inj. Atracurium 0.5 mg/kg — It was given to induce muscle relaxation during anesthesia
Drug: Sevoflurane 2.5 vol % — It was given to maintain anesthesia during surgery alongwith oxygen in air mixture
Drug: Inj. Cefuroxime 1.5 g IV — It was given as prophylactic antibiotic. 2 doses given. 1st 30-60 min before surgery. 2nd 6 hours after surgery
  Other Names: inj. zinacef
Drug: Drug: Inj. Ketorolac 30 mg IV — 3 doses for analgesia. 1st immediate postoperative, 2nd at 8 hours postoperative and 3 rd at 16 hours postoperative period
Drug: Inj. Zantac 50mg IV — 2 doses. 1st at immediate postoperative and 2nd 12 hours after surgery

SUMMARY:
In our study the investigators want to evaluate the effects of EFTs (emotional freedom techniques) for reducing incidence of PONV (Postoperative nausea and vomiting). The effects of EFTs have been quiet evident on many aspects if the incidence of PONV is reduced then it will be much valuable adjunct to postoperative management of the patients.

Our hypothesis was Emotional freedom techniques are very useful to reduce the incidence of postoperative nausea and vomiting after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The laparoscopic cholecystectomy is now considered as the gold standard for gall stone disease worldwide and over 90% of cholecystectomies are now performed laparoscopically. Due to variety of factors, postoperative nausea and vomiting (PONV) which occurs in 40-70 % of patients undergoing laparoscopic cholecystectomy (LC) is sometimes much troublesome to manage. To reduce the incidence of PONV many drugs and modifications were introduced, such as use of dexamethasone, serotonin receptor antagonists, changing drugs and dosages during anesthesia and acupressure. All these measures except acupressure have some degree of side effects on patients.

The Emotional Freedom Techniques (EFTs) which has been pioneered by Gary Craig is a form of alternate medicine which works by tapping on body energy meridian points. Unlike drugs the EFTs has no side effects too. The role of EFTs for various kinds of physical and mental problems has been established and has shown quite significant results. Initially EFTs were used for psychological benefits but later on research proved that it works on the physical and biochemical levels too which is comparable to the various drugs which act by biochemical changes on human body.

In our study we want to evaluate the effects of EFTs for reducing incidence of PONV. The effects of EFTs have been quiet evident on many aspects if the incidence of PONV is reduced then it will be much valuable adjunct to postoperative management of the patients. We have taken into the consideration of PONV only and after promising results we can evaluate EFTs on more and more other aspects of patient management After meeting inclusion and exclusion criteria, All patients were given Tab. Midazolam 7.5 mg PO at night before surgery and received same standard general anesthesia with endotracheal intubation. Inj. Midazolam IV 0.7 mg/kg was given 45 min before surgery as premedication. Anesthesia was induced by propofol (2.5 mg/kg) after 3 minutes of preoxygenation. Muscle relaxation was achieved by atracuium (0.5 mg/kg). Anesthesia was maintained with sevoflurane (2.5 vol %) and oxygen in air mixture (0.50 ratio). Ventilation was controlled mechanically and end tidal normocapnia was maintained by keeping pCO2 at 35-38 mmHg.

Following medications were given to patients during the process.

* Inj. Cefuroxime 1.5 gm. IV (2 doses, 1st dose 30-60 min before surgery and 2nd dose 6 hours after surgery)
* Inj. Ketorolac 30mg IV (3 doses total, 1st dose immediate postop, 2nd and 3rd at 8 and 16 hours after surgery respectively)
* Inj. Zantac 50 mg IV (2 doses total, 1st immediate postop and 2nd at 12 hours after surgery) All patients were operated by the consultant surgeons. After surgery ward all patients received same standard postoperative care. At 6 hour postoperative period all patients were assessed for PONV by VDS. Then patients were divided randomly into two groups equally by consecutive non probability sampling. Group A was control group while Group B received one session of EFTs tapping for 5 to 10 min. All patients were assessed by PONV at 7, 10 and 15 hours postoperatively. Rescue antiemetic (inj. Metoclopramide 10mg IV) was used when the score of PONV was 2 or more on VDS. To see the effectiveness of EFTs in study group the no. of injections of metoclopramide were not counted at 6 hour postoperatively i.e. before intervention of EFTs.

All the data was recorded on specially designed Performa. Statistical analysis: Data was analyzed using SPSS version 12. Mean and standard deviation were calculated for quantitative data like age, frequency of antiemetic injections. Frequency and percentages were calculated for qualitative data like gender, PONV on the basis of VDS scale. The results were finally analyzed and compared for the two groups using Chi-square test and Mann Whitney U tests where applicable. A p value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective laparoscopic cholecystectomy for gallstone disease.
2. Patients with age range of 25 to 55 years

Exclusion Criteria:

1. H/O chronic illness like DM, IHD, CRF, CLD,
2. H/O acute or chronic psychiatric or psychological illness.
3. H/O APD (acid peptic disease) or regurgitation.
4. H/O of any chemotherapy (cancer drugs, opioids), radiotherapy, any history of repeated infection.
5. H/O use of hepatotoxic drugs like acetaminophen, ciprofloxacin, ATT, valproic acid etc. in last one month.
6. H/O alcohol intake in last one month.
7. Previous hepatobilliary surgery.
8. Complicated cholecystectomy in which laparoscopic cholecystectomy is converted to open cholecystectomy.
9. Patients who are given opioids in postoperative period.
10. Patients who need epidural analgesia in postoperative period.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting. | will be measured at upto 15 hours postoperatively.
  Both groups will be assessed for postoperative nausea/vomiting by VDS (verbal descriptive scale) at 6, 7, 10 and 15 hours respectively.
  Verbal descriptive Scale 0 No nausea
  1. Mild nausea
  2. Moderate nausea
  3. Frequent vomiting
  4. Severe vomiting
Rescue antiemetic | It will be measured upto 15 hours postoperatively.
  Both groups will receive rescue antiemetic i.e. inj. Metoclopramide 10mg IV when there will be 2 or more score on VDS (verbal descriptive scale).

OTHER OUTCOMES:
age | age of the patient at study time in years. average was 30 years approximately.
  age of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Fazal H Shah, FCPS I, Principal Investigator — Benazir Bhutto Hospital, Rawalpindi; Aurangzeb Khan, FCPS, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Jahangir S Khan, FCPS, FACS, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Muhammad B Habshi, FCPS I, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Muhammad Z Saeed, FCPS I, Study Chair — Benazir Bhutto Hospital, Rawalpindi; Sheikh F Riaz, FCPS I, Study Chair — Benazir Bhutto Hospital, Rawalpindi
Locations (1):
- Benazir Bhutto Hospital Rawalpindi., Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Background] Eryilmaz HB, Memis D, Sezer A, Inal MT. The effects of different insufflation pressures on liver functions assessed with LiMON on patients undergoing laparoscopic cholecystectomy. ScientificWorldJournal. 2012;2012:172575. doi: 10.1100/2012/172575. Epub 2012 Apr 24. PMID 22619616
- [Background] Feng PH, Chu KS, Lu IC, Shieh JP, Tzeng JI, Ho ST, Wang JJ, Chu CC. Haloperidol plus ondansetron prevents postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy. Acta Anaesthesiol Taiwan. 2009 Mar;47(1):3-9. doi: 10.1016/S1875-4597(09)60013-8. PMID 19318293
- [Background] Bianchin A, De Luca A, Caminiti A. Postoperative vomiting reduction after laparoscopic cholecystectomy with single dose of dexamethasone. Minerva Anestesiol. 2007 Jun;73(6):343-6. PMID 17589423
- [Background] Craig G. The EFT Manual. Available from: http://www.spiritual-web.com/downloads/eftmanual.pdf
- [Background] Church D, De Asis MA, Brooks AJ. Brief group intervention using emotional freedom techniques for depression in college students: a randomized controlled trial. Depress Res Treat. 2012;2012:257172. doi: 10.1155/2012/257172. Epub 2012 Jul 17. PMID 22848802
- [Background] Church D, Hawk C, Brooks AJ, Toukolehto O, Wren M, Dinter I, Stein P. Psychological trauma symptom improvement in veterans using emotional freedom techniques: a randomized controlled trial. J Nerv Ment Dis. 2013 Feb;201(2):153-60. doi: 10.1097/NMD.0b013e31827f6351. PMID 23364126
- [Background] Church D, Yount G, Brooks AJ. The effect of emotional freedom techniques on stress biochemistry: a randomized controlled trial. J Nerv Ment Dis. 2012 Oct;200(10):891-6. doi: 10.1097/NMD.0b013e31826b9fc1. PMID 22986277
- [Background] Stapleton P, Church D, Sheldon T, Porter B, Carlopio C. Depression symptoms improve after successful weight loss with emotional freedom techniques. ISRN Psychiatry. 2013 Jul 28;2013:573532. doi: 10.1155/2013/573532. eCollection 2013. PMID 23984182
- See also: EFTs manual — http://spiritual-web.com/downloads/eftmanual.pdf